CLINICAL TRIAL: NCT05172076
Title: COVID-19-associated Anxiety of Pregnant Women for Anomalies, Stillbirth and Preterm Labor-2
Acronym: CAASP2
Status: Completed | Type: Observational
Sponsor: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Marcus Riemer, MD, Principal Investigator, Martin-Luther-Universität Halle-Wittenberg
Other Study IDs: 2021-228
Record Dates: First submitted 2021-12-25; First posted 2021-12-29 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Anxiety State
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Capture of anxiety for anomalies, stillbirth and preterm labor of pregnant women during COVID-19 pandemia

ELIGIBILITY:
Inclusion Criteria:

* consenting ability

Exclusion Criteria:

* language barrier
* uncompleted questionary

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: pregnant women between 33 until 37 weeks of gestations with planned labor in University Hospital of Halle or St.Elisabeth and St.Barbara Hospital Halle, Germany
Sampling Method: Probability Sample
Enrollment: 276 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
anxiety for anomalies during COVID-19-pandemic and before (percentage difference in agreement to the items of the questionnaire) | 6 months
  Measurement of self-reported anxiety by a questionnaire and State-Trait Anxiety Inventory (STAI) and comparison (cut-off values) with different empiric studies of anxiety for anomalies in pandemics
anxiety for stillbirths during COVID-19-pandemic and before (percentage difference in agreement to the items of the questionnaire) | 6 months
  Measurement of self-reported anxiety by a questionnaire and State-Trait Anxiety Inventory (STAI) and comparison (cut-off values) with different empiric studies of anxiety for stillbirths in pandemics
anxiety for preterm labour during COVID-19-pandemic and before (percentage difference in agreement to the items of the questionnaire) | 6 months
  Measurement of self-reported anxiety by a questionnaire and State-Trait Anxiety Inventory (STAI) and comparison (cut-off values) with different empiric studies of anxiety for preterm labour in pandemics

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - KH St.Elisabeth und St.Barbara, Halle, Saxony-Anhalt
  - University Hospital of Halle, Halle, Saxony-Anhalt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: First Trial CAASP NCT04568551 — https://clinicaltrials.gov/ct2/show/NCT04568551